CLINICAL TRIAL: NCT04050527
Title: International, Multicentre, Observational, Prospective, Longitudinal Study to Assess the Effectiveness of AboBoNT-A Injections for Adult Lower Limb Spasticity in a Real Life Cohort (AboLiSh)
Brief Title: Study to Assess the Effectiveness of AboBoNT-A Injections for Adult Lower Limb Spasticity in a Real Life Cohort
Acronym: AboLiSh
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-FR-52120-255; 2018-004369-15 (EudraCT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-08 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Adult Lower Limb Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the protocol is to assess the longitudinal attainment of person-centered and function related goals of patients who receive AbobotulinumtoxinA (aboBoNT-A) injections for adult lower limb spasticity over a period of 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects ≥18 years of age
* Primary diagnosis with unilateral adult lower limb nonprogressive spasticity.
* Subject able to take more than five steps with or without assistance.
* Decision to treat the lower limb with aboBoNT-A by the care provider made prior to, and independently from, the decision to enroll the subject in the observational study as per country label.
* Previously untreated with BoNT-A (i.e. naïve to BoNT-A), or previously treated with a BoNT-A (i.e. non-naïve to BoNT-A). For those who were previously treated with BoNTA, they should have responded to BoNT-A treatment and at least 12 weeks should have elapsed from prior injection.
* Signed informed consent prior to participation in the study.

Exclusion Criteria:

* Prior history of nonresponsiveness to BoNT-A therapy
* Previous treatment with BoNT-A of less than 12 weeks prior to enrolment in study.
* Current participation in any other clinical study or have participated within the 12 weeks prior to the Inclusion visit (Visit 1) of this study.
* Severe limitations in passive range of motion/contractures in the affected limb (MAS=4 in at least one of the joints in the lower limb).
* Limb surgery or intrathecal baclofen therapy placement for spasticity within 3 months.
* Nonambulatory subject.
* Pregnant and lactating women.
* Progressive neurological conditions or diagnosis of cerebral palsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a primary diagnosis of unilateral adult lower limb nonprogressive focal spasticity
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Subject centred Goal Attainment Scaling Leg T score (GASleg T) | 16 months
  Mean individual GASleg T score. Goal attainment for each goal will be recorded clinically on a 5-point verbal rating scale (range -2 to +2) and goal scores combined to give an aggregated T score using a standard formula (GASleg T score). Range meaning is -2 = much less than expected and +2 = much more than expected.
  The subject and/or caregiver to identify the main goal areas and establish agreed person centred and function related goals guided by GASleg (usually one primary and up to two secondary goals) at each visit. Goal attainment will be evaluated at the routine follow up visit.
  Goals will be redefined and/or newly set at each injection visit or as per routine practice if further injections are not given. Goals will be SMART [Specific, measurable, attainable, relevant, and time-based]

SECONDARY OUTCOMES:
Muscle tone | 16 months
  Muscle tone will be evaluated using the Modified Ashworth Scale (MAS) /Tardieu Scale according to clinical practice. The MAS is a six point scale (with available scores of 0, 1, 1+, 2, 3 and 4) reporting changes in muscle tone during muscle flexion or extension. Tardieu scale quantifies muscle spasticity by assessing the response of the muscle to stretch applied at specified velocities. It can therefore broadly differentiate between the two key factors explaining resistance to passive stretch, namely contracture (non-neural factors) and spasticity (neural factors).
Severity of different aspects of impairment | 16 months
  Severity of different aspects of impairment in subjects with neurological injury will be evaluated using the Lower Limb Spasticity adapted Neurological Impairment Scale. (LLS-NIS) Higher LLS-NIS scores indicate more severe impairment (LLS-NIS). Higher LLS-NIS scores indicate more severe impairment.
Total dose injected per cycle | 16 months
Report muscles injected | 16 months
Report dose per muscle | 16 months
Assess correlations of subject centered goals | 16 months
  Correlations of subject centred goals and related standardised rating scales will be assessed using GASleg and standardised outcome measures selected according to the goals for treatment.
Evolution of Quality of Life | 16 months
  Assess the evolution of QoL at each visit based on the EQ-5D-5L and the QoL element of LegA. This is a descriptive scale that covers 5 dimensions: mobility, self-care, usual activities,pain/discomfort and anxiety/depression. the scale consist of 5 levels, where level one corresponds to "no problems" and level 5 corresponds to "extreme problem".

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (51):
- United States (16):
  - Rancho Los Amigos National Rehabilitation Center (RLANRC) - Neurology, Downey, California
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Kansas City Bone and Joint Clinic, P.A. (KCBJ) - Overland Pa, Leawood, Kansas
  - Neurology Center of NE,PC - Neurology, Foxborough, Massachusetts
  - Beaumont Hospital, Grosse Pointe - Neurology, Grosse Pointe, Michigan
  - Yeshiva University - Albert Einstein College of Medicine - Montefiore Medical Center (MMC) - Neurology, The Bronx, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Riverhills Healthcare, Cincinnati, Ohio
  - OrthoNeuro, Columbus, Ohio
  - Good Shepherd Rehabilitation Hospital - Neurology, Allentown, Pennsylvania
  - MossRehab - Einstein Medical Center, Elkins Park, Pennsylvania
  - Rehabilitation Associates - Neurology, Paoli, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - The University of Utah School of Medicine, Salt Lake City, Utah
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (2):
  - Princess Alexandra Hospital, Ipswich
  - Royal Prince Alfred Hospital, Rozelle
- Brazil (2):
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto (HCFMRP) - Neurology, Ribeirão Preto
  - Hospital de Base de São José do Rio Preto at Centro Integrado de Pesquisa (CIP) - Neurology, São José do Rio Preto
- Canada (3):
  - Glenrose Rehabilitation Hospital, Edmonton
  - River Valley Health - Stan Cassidy Foundation - Stan Cassidy, Fredericton
  - McGill University Health Center, Montreal
- France (6):
  - CHU - HÃ´pital Pellegrin - Neurologie, Bordeau
  - CHU RAYMOND POINCARE - Neurology, Garches
  - Centre Hospitalier Regional Universitaire (CHRU) de Lille - Hopital Pierre Swynghedauw - Neurology, Lille
  - Höpital Sainte-Marie - Neurology, Paris
  - Centre Hospitalier Universitaire De Reims - Hopital Maison B, Reims
  - Pole Saint Helier, Rennes
- Germany (5):
  - Neurologie und Psychosomatik am Wittenbergplatz, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Medizinische Hochschule Hannover - Neurology Neurologische Poliklinik, Hanover
  - Universitätsklinikum/Neurologie, Lübeck
  - Neurologische Klinik und Poliklinik, Würzburg
- Italy (5):
  - Università Degli studi della Campania - Luigi Vanvitelli - Neurologica, Napoli
  - Istituto Scientifico di Riabilitazione di Veruno, Fondazione, Novara
  - PO Villa Sofia, AO Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - AO S.Camillo-Forlanini, Roma
  - Universita degli Studi di Verona - Centro di Ricerca in Riabilitazione Neuromotoria e Cognitiva (CRRNC) - Neurology, Verona
- Poland (5):
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Wojew. Wielospecjalistyczne Centrum Onkologii i Traumatologii im.M.Kopernika w Lodzi, Lodz
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Mazowiecki Szpital Brodnowski w Warszawie Sp. z o.o. Brodnowskie Centrum Kliniczne Poliklinika Brodnowskiego Centrum Klinicznego, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
- Russia (7):
  - Regional state budget health institution "City Hospital № 5", Barnaul
  - SAHI Interregional Clinical Diagnostic Center, Kazan'
  - National Medical Research Treatment and Rehabilitation Center of the Ministry of Health of Russia, Moscow
  - Bekhterev National Research Medical Center for Psychiatry, Saint Petersburg
  - Pavlov First Saint-Petersburg State Medical University - Neurology, Saint Petersburg
  - Federal State Budgetary Institution "All-Russian Center for Emergency Medicine and Medical Radiology named after A.M. Nikiforov" of the EMERCOM of Russia, Saint Petersburg
  - FGBOU VO "Ural state medical university", Yekaterinburg

REFERENCES:
- [Derived] Esquenazi A, Zorowitz RD, Ashford S, Jacinto J, Beneteau M, Maisonobe P, Hannes C, Sandars S. Achieving treatment goals with repeated injections of botulinum toxin in adults with leg spasticity. Curr Med Res Opin. 2025 Dec 25:1-9. doi: 10.1080/03007995.2025.2606555. Online ahead of print. PMID 41449804
- [Derived] Esquenazi A, Zorowitz RD, Ashford S, Beneteau M, Maisonobe P, Hannes C, Jacinto J; AboLiSh Study Group. Longitudinal Goal Attainment With Repeat Injections of AbobotulinumtoxinA in Adults With Lower Limb Spasticity: Results From a Prospective Observational Study. Arch Phys Med Rehabil. 2025 Jun;106(6):894-901. doi: 10.1016/j.apmr.2024.10.017. Epub 2024 Nov 20. PMID 39571744
- [Derived] Esquenazi A, Zorowitz RD, Ashford S, Maisonobe P, Page S, Jacinto J. Clinical presentation of patients with lower limb spasticity undergoing routine treatment with botulinum toxin: baseline findings from an international observational study. J Rehabil Med. 2023 Oct 5;55:jrm4257. doi: 10.2340/jrm.v55.4257. PMID 37794845